CLINICAL TRIAL: NCT06953713
Title: Umbilical Trochar Site Is The Usual Suspect For Trocar Hernia After Laparoscopic Cholecystectomy: A Prospective Study
Brief Title: TSH Risk by Extraction Site in Lap Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Basak (Other Government)
Responsible Party: Sponsor-Investigator, Fatih Basak, Professor, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/27
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Gallstone
Keywords: Trocar site hernia; laparoscopic cholecystectomy; incisional hernia; port site hernia
MeSH Terms: conditions — Gallstones; Incisional Hernia

STUDY DESIGN:
Intervention Model Description: A standard four-trocar LC was performed using a 10 mm umbilical camera trocar, a 10 mm epigastric trocar, and two 5 mm subcostal trocars. The gallbladder was retrieved using a laparoscopic specimen bag through either:
  Group U: Gallbladder retrieved via the umbilical trocar, Group E: Gallbladder retrieved via the epigastric trocar.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical group (Group U) (Experimental): Gallbladder retrieved via the umbilical trocar following standard 4-port laparoscopic cholecystectomy
  Interventions: Procedure: gallbladder extraction umbilical
- Epigastric group (Group E) (Active Comparator): Gallbladder retrieved via the epigastric trocar following standard 4-port laparoscopic cholecystectomy
  Interventions: Procedure: extracting gallbladder via epigastric port

INTERVENTIONS:
Procedure: gallbladder extraction umbilical — extracting gallbladder via umbilical port site
  Arms: Umbilical group (Group U)
Procedure: extracting gallbladder via epigastric port — extracting gallbladder via epigastric port
  Arms: Epigastric group (Group E)

SUMMARY:
The main purpose of this study is to determine whether removing the gallbladder through different incision sites (ports) during laparoscopic surgery affects the risk of developing an incisional hernia. All patients undergo the same number of incisions, and the surgical technique remains standardized.

The study also aims to identify other factors that may contribute to the risk of hernia formation following gallbladder surgery.

DETAILED DESCRIPTION:
Patients were blinded to group assignment. Randomization was conducted on the day of surgery by a surgical nurse using the Alea Randomisation mobile application (Alea Clinical Services, Abcoude, Netherlands). Group allocation ("U" for umbilical or "E" for epigastric) was placed in a sealed envelope and delivered to the operating room. The envelope was opened by the attending surgeon immediately prior to gallbladder retrieval.

Due to the nature of the intervention, the operating surgeon could not be blinded; however, surgeons remained unaware of group allocation until the moment of specimen retrieval. All procedures were performed by one of three experienced surgeons.

A conventional four-port laparoscopic cholecystectomy was performed in all cases, using a 10 mm umbilical camera trocar, a 10 mm epigastric trocar, and two 5 mm subcostal trocars. Gallbladder retrieval was performed using a laparoscopic specimen bag through one of the following approaches:

Group U: Gallbladder retrieved through the umbilical trocar

Group E: Gallbladder retrieved through the epigastric trocar

After retrieval and hemostasis, all trocars were removed under direct laparoscopic vision. The umbilical fascia was closed using two interrupted polyglactin 910 sutures (Vicryl, Ethicon Inc., Edinburgh, Scotland), while the epigastric trocar fascia was left unsutured. Fascia closure practices were standardized and unrelated to group allocation. Total operation time and gallbladder retrieval time were recorded.

All patients received paracetamol (Parol, Atabay İlaç, Istanbul, Türkiye) three times daily and tramadol (Contramal, Abdi İbrahim İlaç, Istanbul, Türkiye) twice daily for postoperative pain control. Pain was assessed using the Visual Analogue Scale (VAS) at 6 and 24 hours postoperatively, with the assistance of a ward nurse.

Patients without complications were discharged on postoperative day 1. Those with complications were discharged following resolution of their condition. All patients were followed for one year postoperatively. Patients presenting with hernia-related symptoms (e.g., bulge or pain) underwent ultrasonography (USG) at symptom onset, while asymptomatic patients received routine USG at the six-month and one-year follow-ups. Radiologists performing USGs were not affiliated with the study and were not standardized.

Incisional hernia was defined as a pathological fascial defect at a postoperative trocar site with protrusion of intraabdominal contents. Both clinically and radiologically diagnosed hernias were considered incisional hernias.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Gallbladder stones
* No known systemic comorbidities (e.g., cardiovascular, pulmonary, metabolic, or immunologic conditions)

Exclusion Criteria:

* Age < 18 years,
* Open cholecystectomy or conversion from laparoscopy to open surgery,
* Acute cholecystitis
* Prior intervention involving the common bile duct,
* Presence of clinical or radiologic diastasis recti,
* Presence of clinical or radiologic umbilical hernia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Trocar Site Hernia Following Laparoscopic Cholecystectomy | From operation to end of follow-up period at 1 year
  The primary outcome is to determine whether the site of gallbladder retrieval influences the incidence of postoperative incisional hernia following laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Postoperative Pain Assessed by Visual Analog Scale (VAS) at 6 and 24 Hours | From end of operation to postoperative 24 hours
  This outcome evaluates the relationship between the gallbladder extraction site and postoperative pain, measured using the Visual Analog Scale (VAS) at 6 and 24 hours after surgery. The VAS is a 10-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain severity.
Incidence of Trocar Site Hernia in Relation to Patient- and Surgery-Related Risk Factors | From operation to end of follow-up period at 1 year
  This outcome measures the incidence of trocar site hernia during a one-year follow-up and evaluates its statistical correlation with various clinical and surgical risk factors. These include age (years), sex (male/female), BMI (kg/m²), diabetes status (yes/no), extraction site location (umbilical or epigastric), fascial closure status (closed/open), and intraoperative widening of the extraction site (yes/no). The hernia diagnosis will be based on clinical evaluation and ultrasonographic confirmation.
  Data will be analyzed using correlation or regression methods to assess the strength of association between these variables and hernia development.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Research and Training Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Raw data, consent forms, CSR, SAP
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Unending (e.g., "Beginning 1 year after publication with no end date")
Access Criteria: Statistical methods for those analyses must be approved by independent review. A proposal that describes planned analyses must be submitted
URL: https://osf.io/q9yga/?view_only=3918142092a9459fa1f4a96ebae6811b

REFERENCES:
- [Background] Sood S, Imsirovic A, Sains P, Singh KK, Sajid MS. Epigastric port retrieval of the gallbladder following laparoscopic cholecystectomy is associated with the reduced risk of port site infection and port site incisional hernia: An updated meta-analysis of randomized controlled trials. Ann Med Surg (Lond). 2020 May 25;55:244-251. doi: 10.1016/j.amsu.2020.05.017. eCollection 2020 Jul. PMID 32528673

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT06953713/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT06953713/ICF_001.pdf